CLINICAL TRIAL: NCT00476853
Title: A 48 Week, Randomized, Open-label, 2 Arm Study to Compare the Efficacy, Safety and Tolerability of HAART Containing Nevirapine 400mg/Day Versus Nevirapine 600 mg/Day in HIV-1 Infected Patients Started at 2-6 Weeks After Initiating Rifampin Containing Antituberculous Therapy
Brief Title: Efficacy Safety Study Comparing 2 Doses of NVP After Initiating Rifampin-containing TB Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: other sponsors:Japanese MOPH (Unknown); Labor and Welfare (Unknown); Thai MOPH (Unknown); Thai GPO (Unknown); Bamrasnaradura Infectious Diseases Institute (Other Government); Chiang Rai Hospital (Other); King Chulalongkorn Memorial Hospital (Other); Central General Chest Institute (Unknown); The Research Institute of Tuberculosis (Japan) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 033
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV-TB; nevirapine based HAART with rifampin treated TB; Compare PK profile, efficacy, safety and tolerability of HAART containing nevirapine 400mg/day versus 600 mg/day in HIV/TB co-infected patients; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): NVP 400 mg
  Interventions: Drug: HAART containing nevirapine
- 2 (Active Comparator): NVP 600 mg
  Interventions: Drug: HAART containing nevirapine

INTERVENTIONS:
Drug: HAART containing nevirapine — Initially NVP 200 mg BID (400 mg per day) was compared to 400 mg BID and 200 mg OD NVP (600 mg per day). 400 mg/day versus 600 mg/day.

SUMMARY:
A 48 week, randomized, open-label, two arm study to compare the efficacy, safety and tolerability of HAART containing nevirapine 400 mg/day versus nevirapine 600 mg/day in HIV-1 infected patients started at 2-6 weeks after initiating rifampicin containing antituberculosis therapy.

DETAILED DESCRIPTION:
Preliminary data from the HIVNAT PK laboratory indicate that out of 5/60 patients treated with nevirapine (200 mg bid) and rifampicin had sub-therapeutic nevirapine levels (<3.0 mg mg/L). In a control group of 38 patients using nevirapine without rifampicin there were no sub-therapeutic levels. A dose increase of nevirapine while patients who are receiving that rifampicin may be required. Both nevirapine and rifampicin are tepatotoxic agents as are other agents used in treatment of HIV or tuberculosis. Using a higher nevirapine may prevent the occurrence of sub-therapeutic nevirapine levels, but may also induce more liver toxicity. To address these issues, we designed a randomized prospective study to evaluate the safety, efficacy and pharmacokinetics of nevirapine 400 mg/day versus 600 mg/day with a two weeks lead-in 200 mg/day and 400 mg/day respectively, in TB-HIV co-infected patients who taking rifampicin and short-term efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV positive after voluntary counseling and testing
2. Aged 18-60 years of age
3. Antiretroviral treatment naïve.
4. CD4+ cell count of < 200 cells/mm3 at the time of diagnosed TB
5. TB is diagnosed and using treatment with rifampin base therapy for at least 2 weeks but no longer than 4 weeks duration. The requirement for study entry is at least one acid-fast bacillus (AFB) positive smear with a typical syndrome and/or CXR findings consistent with pulmonary TB. Pulmonary TB and / or extra pulmonary TB will be included if AFB or culture for TB is positive.
6. No other active OI (CDC class C event)
7. Negative pregnancy test in females, and willing to use reliable contraception
8. Able to provide written informed consent.

Exclusion Criteria:

1. The following laboratory variables, i. absolute neutrophil count (ANC) < 1000 cells/uL ii. hemoglobin < 6.5 g/dL iii. platelet count < 50,000 cells/uL iv. serum AST, ALT > 5 x ULN vi. serum bilirubin > 2 x ULN vii. serum creatinine > 2 x ULN viii. Pregnant or nursing mothers.
2. Current use of steroid and other immunosuppressive agents.
3. Current use of any prohibited medications related to compliance and drug pharmacokinetics (see appendix )
4. Acute therapy for serious infection or other serious medical illness (in the judgment of the site Principal Investigator) requiring systemic treatment and/or hospitalization.
5. Patients with current alcohol or illicit substance use that in the opinion of the site Principal Investigator would conflict with any aspect of the conduct of the trial.
6. The persons who had been received a mono-therapy of nevirapine
7. Unlikely to be able to remain in follow-up for the protocol defined period.
8. Patients with chronic active liver disease.
9. Patients with proven or suspected acute hepatitis. Patients with chronic viral hepatitis are eligible provided ALT, AST < 5 x ULN.
10. Karnofsky performance score <30%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of nevirapine based HAART 400 mg/day versus 600 mg/day on HIV-1 load as measured by HIV-1 RNA quantification in plasma | 48 weeks

SECONDARY OUTCOMES:
Safety and tolerability of nevirapine based HAART 400 mg/day versus 600 mg/day | 48 weeks
Nevirapine level at week 2, 4 and 12 and 12 hour PK at week 4 (only 20 patients) | 48 weeks
Immune recovery syndrome, adherence, clinical improvement, incidence of new/recurrent AIDS events (CDC class C) between two group | 48 weeks
Time to mortality or new/recurrent AIDS events (CDC class C), 1 year mortality rate of TB/HIV patients, emerging of ARV resistant especially nevirapine, emerging of anti-TB resistance | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)
Locations (6):
- Thailand (6):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Chiangrai Hospital, Chiang Rai
  - Mae Chan Hospital, Chiang Rai
  - Phan Hospital, Chiang Rai
  - Bamrasnaradura Institute, Nonthaburi
  - Central Chest Hospital, Nonthaburi

REFERENCES:
- [Derived] Avihingsanon A, Manosuthi W, Kantipong P, Chuchotaworn C, Moolphate S, Sakornjun W, Gorowara M, Yamada N, Yanai H, Mitarai S, Ishikawa N, Cooper DA, Phanuphak P, Burger D, Ruxrungtham K. Pharmacokinetics and 48-week efficacy of nevirapine: 400 mg versus 600 mg per day in HIV-tuberculosis coinfection receiving rifampicin. Antivir Ther. 2008;13(4):529-36. PMID 18672531
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org